CLINICAL TRIAL: NCT06782399
Title: A Pilot of a Microdevice for in Situ Candidate Drug Screening of Cutaneous Lesions of Squamous Cell Carcinoma
Brief Title: Drug Screening of Cutaneous Lesions of Squamous Cell Carcinoma
Acronym: SCC
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oliver Jonas (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Oliver Jonas, Associate Professor, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-379
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Squamous Cell Carcinoma of the Skin; Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Skin; Implantable Microdevice
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local treatment cohort (Experimental): Local Treatment Cohort (5 participants) may recruit participants who plan to receive local surgical intervention (Mohs surgery or local excision) alone or in combination with further surgical treatment, radiation, or systemic therapy.
  Interventions: Combination Product: Microdevice
- Systemic treatment cohort (Experimental): Systemic Treatment Cohort (20 patients) will not enroll until initial cohort has been completed (MD have been implanted, retrieved, and processed for immunohistochemical analysis). Microdevice protocol will be optimized given results derived from the local treatment cohort. Will include participants who plan to receive systemic therapy in the absence of additional local therapy (surgery or radiation). If patients receive systemic therapy, and there is clinical cutaneous residual disease after 12 weeks of systemic therapy, an additional 1 to 4 MDs will be implanted into residual cutaneous disease at this time.
  Interventions: Combination Product: Microdevice

INTERVENTIONS:
Combination Product: Microdevice — Device: Microdevices
  The microdevice is an investigational miniaturized implantable nanodose drug delivery device. It was developed as a tool with the ultimate goal to help screen several existing and investigational drugs directly within a patient's tumor to identify what drugs are the most effective for treating a patient's cancer. The microdevice releases nanodoses of several approved drugs into the tumor, and is then excised minimally invasively several days later.
  Other: Standard of care therapy
  Participant to receive standard of care therapy as previously determined by participant's treating oncologist and/or dermatologist, which may include a skin-directed or systemic therapy

SUMMARY:
This research study is studying the effect of different drugs as possible treatments for squamous cell carcinoma (SCC).

DETAILED DESCRIPTION:
The pilot study will determine the feasibility of using an in situ microdevice to measure local intratumoral response to several cancer treatments in patients with cutaneous lesions of squamous cell carcinoma.

This research study is a Pilot Study, which is the first-time investigators are examining this study device in SCC. The treatment received will be the normal standard-of-care treatment for SCC However, the placement and removal of the microdevice is being tested for the first time in this type of cancer.

This research study involves drugs that are released by a small implantable microdevice (IMD) as small as the tip of a needle, that is inserted into the tumor and is then removed 3-5 days later. The microdevice can hold up to 20 drugs in very small concentrations that are able to access the cancer through small pores in the device. When the device is removed along with the cancer 3-5 days later, it will be evaluated to understand which drug(s) may be effective to treat these cancers.

The U.S. Food and Drug Administration (FDA) has not approved the microdevice a treatment for any disease.

AACRF, a research foundation, is supporting this research study by providing funding for the research study, the study drugs and study procedures

ELIGIBILITY:
Inclusion Criteria:

* Participants must have clinical diagnosis of cutaneous squamous cell carcinoma or metastatic squamous cell carcinoma with cutaneous involvement supported by histological evaluation of skin lesions based upon available clinical data including pathology reports from non-study institution (if applicable)
* Participants must have visible cutaneous disease. Skin lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* A single lesion is amenable to placement of one or multiple devices in terms of lesion size and location, as assessed by dermatologist (minimum lesion diameter of 1.0 cm).
* Washout period from previous treatments is not necessary.
* Age minimum of age 18. Because of limited incidence of cutaneous squamous cell carcinoma in the pediatric population, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Participants will undergo laboratory testing within 28 days prior to the procedure. Participants must have marrow function as defined below:

absolute neutrophil count ≥500/mcL platelets ≥50,000/mcL

* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the efficacy assessment of the systemic regimen are eligible for this trial in the systemic treatment cohort (expansion cohort).
* Participants must be evaluated by a dermatologist or medical oncologist who will determine the clinically appropriate treatment strategy based on clinical history and extent of disease. Systemic therapy will be mandatory for expansion/systemic treatment cohort. Systemic therapy may be initiated anytime within 4 weeks of MD removal.
* Patients must be deemed medically stable to undergo percutaneous procedures by their treating cutaneous oncologist.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must be willing to undergo research-related genetic and transcriptomic sequencing (somatic and germline) and data management, including the deposition of de-identified genetic sequencing data in NIH central data repositories.
* Patient is considered to have capacity to properly follow instructions at home for the care of device(s) (see Appendix B).

Exclusion Criteria:

* Positive serum pregnancy test at screening visit. Pregnant women are excluded from this study because the agents used for microdosing have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is enrolled in this study.
* Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or biopsy procedures.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who will receive standard of care systemic therapy in expansion cohort are not allowed to start any new skin directed therapy (e.g. topical 5-fluorouracil, imiquimod, etc.) concurrent with first systemic therapy initiated after device implantation and retrieval. Should a patient clinically progress on first systemic therapy and require a change in treatment, skin directed therapies may be introduced if desired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of analysis | through study completion, an average of 1 year
  For the feasibility endpoint, a "successful" procedure will be defined as the ability to retrieve the device (by either skin punch biopsy tool or surgical excision) without damaging tumor tissue surrounding the microdevice, and with a rim of tissue of at least 500um thickness surrounding the microdevice, to allow for downstream immunohistochemistry analysis. At least 80% of the device reservoirs need to be surrounded by tissue in order to be considered successful.
  For purposes of this endpoint, feasibility will be assessed on a per-device basis rather than a per-patient basis, with each device considered relatively independent in terms of placement, retrieval, and analysis.
Cell death index measurement | through study completion, an average of 1 year
  To identify which microdosed targeted or chemotherapeutic cancer agents, delivered by an implantable microdevice in cutaneous lesions of squamous cell carcinoma in the expansion cohort, induce a cell death index value of at least 30% based on quantitative histopathologic assessment.
  To identify which microdosed targeted or chemotherapeutic cancer agents, delivered by an implantable microdevice in cutaneous lesions of squamous cell carcinoma in the expansion cohort, induce a cell death index value of at least 30% based on quantitative histopathologic assessment.
  To identify which microdosed targeted or chemotherapeutic cancer agents, delivered by an implantable microdevice in cutaneous lesions of squamous cell carcinoma in the expansion cohort, induce a cell death index value of at least 30% based on quantitative histopathologic assessment.

SECONDARY OUTCOMES:
Safety | through study completion, an average of 1 year
  To evaluate the safety of microdevice placement and removal based on assessment of adverse events.
Correlation between tumor-drug response on microdevice and clinical response to systemic treatment | through study completion, an average of 1 year
  We will perform a preliminary assessment of the statistical correlation between the extent of tumor response to drug with the microdevice (measured using immunohistochemical analysis of drug-exposed tumor tissue for markers of apoptosis and cell proliferation) and the clinical responses to systemic therapy (via disease measurements including clinical and/or radiographic evidence of disease response).
Additional biomarker identification | through study completion, an average of 1 year
  Immune infiltrates in the local tumor tissue exposed to microdevice delivered drugs.
Intralesional heterogeneity assessment | through study completion, an average of 1 year
  To assess intralesional heterogeneity in drug response by comparing the extent of tumor response to drug among different locations in a single tumor with multiple microdevices.

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu